CLINICAL TRIAL: NCT05147922
Title: Neo RQI: Evaluating the Effect of Neonatal Resuscitation Quality Improvement Cart Booster Training on Provider Positive Pressure Ventilation Skills Retention
Brief Title: Neo RQI: The Effect of Neonatal Resuscitation Quality Improvement Cart Booster Training Skills Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Academy of Pediatrics (Other)
Responsible Party: Principal Investigator, Vishal Kapadia, Associate Professor- Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU2021-0282
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Ventilatory Failure
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Booster Training Group (Experimental): Participants randomized to intervention will undergo booster training sessions with the RQI cart (including audiovisual feedback) at 3, 6 and 9 months post instructor-led training session. Following each of these booster sessions, the participants will undergo 1 minute assessments, without feedback.
  Interventions: Behavioral: Booster Training with the Neonatal Resuscitation Quality Improvement Cart
- No Booster Training Group (No Intervention): Participants randomized to the control group will undergo 1 minute assessments, without feedback, at 6 and 9 months. Participants will not be able to access the RQI cart outside of their assessment.

INTERVENTIONS:
Behavioral: Booster Training with the Neonatal Resuscitation Quality Improvement Cart — The cart will give providers audio-visual feedback and walk them through how to perform effective positive pressure ventilation with correct head positioning, appropriate Peak Inspiratory Pressure and Peak End Expiratory Pressure, no mask leak and ventilation rate of 40 per minute. Participants will be able to spend up to 30 minutes with the cart before undergoing their 1 minute assessment, which will be without feedback.
  Arms: Booster Training Group

SUMMARY:
This is a prospective multicenter randomized control trial to assess percentage mask leak six months post instructor led positive pressure ventilation skills training in providers who undergo booster training compared to those who do not undergo any booster training

DETAILED DESCRIPTION:
Baseline positive pressure ventilation skill assessment of all study participants: Site principal investigators will recruit eligible providers for the trial. Participants will fill out study enrollment sheet which will ask for 1. Demographic information 2. Profession 3. Experience (number of times positive pressure ventilation performed on a newborn in the last 6 months) 4. Last time Neonatal Resuscitation Program course attended and 5. Institution. Participants will perform 1 minute of positive pressure ventilation on the cart. During this baseline assessment, there is no audio-visual feedback or display. The cart will record data on mask leak, pressure used, ventilation rate, head positioning.

Pre-randomization Standardized Instructor Led Skills Training: All study participants will undergo the standard instructor-led positive pressure ventilation skills training. Each site will have a designated study instructor who will remain blinded to the baseline positive pressure ventilation skill assessment data. Study instructors will use a standardized script as a guide for the instructor led positive pressure ventilation skills training. This training will occur with the same manikin and equipment as the one available at the cart. This training will decrease the impact of variability in prior training received by the study participants.

Post- Instructor led positive pressure ventilation skills training Assessment: Immediately after the instructor led training, participants will perform 1-minute positive pressure ventilation on the cart. This will also be a blinded assessment without any display or feedback. Comparison of pre- and post- instructor led training assessments will provide unique data to evaluate if instructor led training changes the positive pressure ventilation skills.

Randomization with minimization procedure: Randomization will be provided by a secure website using the computer-generated randomization and the minimization procedure. The goal of the minimization procedure is to prevent an imbalance of factors that may influence positive pressure ventilation skill retention. Factors that will be taken into account during minimization procedure are

1. PPV skill proficiency during baseline pre-instructor led training assessment: Based on the pre-training skill assessment, each participant will be coded as a Group A [Proficient] or Group B [not proficient]. Participants will be considered proficient if participants are able to achieve low mask leak (< 30%) on >80% of ventilations provided. Only study Principal investigator and research nurse will have access to this data. 2. Profession 3. Experience (number of times positive pressure ventilation performed on a newborn in the last 6 months) 4. Last time NRP course attended and 5. Institution. Based on this information, the randomization website will assign them to the intervention (booster training) or control group (no booster training) with 1:1 allocation.

ELIGIBILITY:
Inclusion Criteria:

* Any Neonatal Resuscitation Program-card carrying provider at the participating sites (University of Texas Southwestern, Stanford University and St. Louis University).

Exclusion Criteria:

* Novice providers, who have never taken an Neonatal Resuscitation Program course, will be excluded as participant may not be familiar with the equipment to initiate positive pressure ventilation skills without a face-to-face interaction with an instructor

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mask Leak | 6 months after initial enrollment and instructor-led training session
  The primary outcome of the study is the proportion of subjects who provide >80% ventilation with low mask leak (< 30% mask leak) during the one-minute assessment at six months from the instructor led positive pressure ventilation skills training

SECONDARY OUTCOMES:
Tidal volumes | 6 month and 9 month assessments
  Measured percentage of breaths provided in goal range for tidal volume
Positive Pressure Ventilation composite score | 6 month and 9 month assessments
  Calculated score, based on peak inspiratory pressure score, positive end expiratory pressure score, rate score, and mask leak score, per provider at each assessment
Peak Inspiratory Pressure score | 6 month and 9 month assessments
  Measured percentage of breaths provided in goal range for peak inspiratory pressure
Positive End Expiratory Pressure score | 6 month and 9 month assessments
  Measured percentage of breaths provided in goal range for positive end expiratory pressure
Rate score | 6 month and 9 month assessments
  Measured percentage of breaths provided in goal range for rate

CONTACTS AND LOCATIONS:
Overall Officials: Priya Sharma, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas, Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wyckoff MH, Wyllie J, Aziz K, de Almeida MF, Fabres J, Fawke J, Guinsburg R, Hosono S, Isayama T, Kapadia VS, Kim HS, Liley HG, McKinlay CJD, Mildenhall L, Perlman JM, Rabi Y, Roehr CC, Schmolzer GM, Szyld E, Trevisanuto D, Velaphi S, Weiner GM; Neonatal Life Support Collaborators. Neonatal Life Support: 2020 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2020 Oct 20;142(16_suppl_1):S185-S221. doi: 10.1161/CIR.0000000000000895. Epub 2020 Oct 21. PMID 33084392
- [Background] Schmolzer GM, Dawson JA, Kamlin CO, O'Donnell CP, Morley CJ, Davis PG. Airway obstruction and gas leak during mask ventilation of preterm infants in the delivery room. Arch Dis Child Fetal Neonatal Ed. 2011 Jul;96(4):F254-7. doi: 10.1136/adc.2010.191171. Epub 2010 Nov 16. PMID 21081593
- [Background] Schmolzer GM, Kamlin OC, O'Donnell CP, Dawson JA, Morley CJ, Davis PG. Assessment of tidal volume and gas leak during mask ventilation of preterm infants in the delivery room. Arch Dis Child Fetal Neonatal Ed. 2010 Nov;95(6):F393-7. doi: 10.1136/adc.2009.174003. Epub 2010 Jun 14. PMID 20547584
- [Background] Martin P, Theobald P, Kemp A, Maguire S, Maconochie I, Jones M. Real-time feedback can improve infant manikin cardiopulmonary resuscitation by up to 79%--a randomised controlled trial. Resuscitation. 2013 Aug;84(8):1125-30. doi: 10.1016/j.resuscitation.2013.03.029. Epub 2013 Apr 6. PMID 23571117